CLINICAL TRIAL: NCT02878239
Title: The Relationship Between the Imaging Assessment Based on Kellgren-Lawrence Scores and In Vivo 3D Knee Kinematic Characteristics in Chinese Patients With Medial Knee Osteoarthritis During Walking Using a New Portal Gait System.
Brief Title: The Three-dimensional Gait Analysis of Medial Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Collaborators: Medical Center of Assessment, Prevention and Treatment of Bone & Joint Diseases, Guangdong, China (Other); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Yu Zhang, chief surgeon, associate professor, Guangzhou General Hospital of Guangzhou Military Command
Other Study IDs: GuangzhouGH001
Record Dates: First submitted 2016-08-16; First posted 2016-08-25 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis
Keywords: knee osteoarthritis; gait; Kellgren-Lawrence Scores
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Early OA: All patients (>35 years) have been diagnosed with medial knee osteoarthritis according to the American College of Rheumatology criteria. Those are classified as patients with early knee osteoarthritis because their Kellgren-Lawrence Scores were Grade I.
  Interventions: Other: Steps 1
- Moderate OA: All patients (>35 years) have been diagnosed with medial knee osteoarthritis according to the American College of Rheumatology criteria. Those are classified as patients with moderate knee osteoarthritis because their Kellgren-Lawrence Scores were Grade II.
  Interventions: Other: Steps 1
- Severe OA: All patients (>35 years) have been diagnosed with medial knee osteoarthritis according to the American College of Rheumatology criteria. Those are classified as patients with moderate knee osteoarthritis because their Kellgren-Lawrence Scores were Grade III/IV.
  Interventions: Other: Steps 1
- Asymptomatic Participants: The asymptomatic participants（>35 years） has no history of knee pain, trauma, surgery, or obvious gait abnormalities. They are set as controls in the study.
  Interventions: Other: Steps 2

INTERVENTIONS:
Other: Steps 1 — Kinematic characteristics are obtained by the portal gait analysis system in the patients. Kellgren-Lawrence Scores are obtained according to their radiography.
  Groups: Early OA; Moderate OA; Severe OA
Other: Steps 2 — Kinematic characteristics are obtained by the portal gait analysis system in the subjects.Physical examinations are taken to avoid other diseases.
  Groups: Asymptomatic Participants

SUMMARY:
Static imaging has been commonly and clinically accepted to assess the severity of medial knee osteoarthritis (KOA), especially the radiography. Gait analysis has been adopted to evaluate the kinematic characteristics of the knees in patients with KOA. Most of the current studies focus on the sagittal plane of the knee, but very few of them focus on the frontal or horizontal plane. With the different severity of medial KOA, anatomical structures of the knees will change and influence kinematics of the knees, such as osteophytes and deformity. At present, there has been no study focusing on the relations between the imaging assessment of the severity and quantitative kinematics of medial KOA. The aim of the study is to explore the relationship between the imaging assessment based on the Kellgren-Lawrence Scores and in vivo 3D knee kinematic characteristics in Chinese patients with medial KOA during walking using a new portal gait system.

DETAILED DESCRIPTION:
All patients are assessed according to the Kellgren-Lawrence Score.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of medial knee osteoarthritis according to the American College of Rheumatology criteria.
2. The patients are confirmed by radiographic evidence that medial tibiofemoral joint space grade was narrower than lateral tibiofemoral joint space.
3. The patients have clinical symptom of medial pain of the knee.
4. Clinical examinations are taken to examine the asymptomatic subjects to avoid knee diseases.

Exclusion Criteria:

1. Traumatic knee osteoarthritis.
2. Lateral tibiofemoral KOA or any other types of Knee OA.
3. Ambiguity of Kellgren-Lawrence scores
4. History of surgery.
5. Neuromuscular disease, cardiovascular disease or trauma that can affects gait.
6. Body mass index greater than 35.
7. Needing stick or assistance to walk or unable to walk at a speed of less than 2.0 km/h and less than 300 m.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese patients diagnosed with medial KOA andasymptomatic participants will be recruited. The asymptomatic participants（>35 years） have no history of knee pain, trauma, surgery, or obvious gait abnormalities.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2016-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Kinematic characteristics of the the six-degree-of-motion (6DOF) of the gait at heel strike in asymptomatic participants and patients with knee osteoarthritis. | 1 Day
  The 6DOF include flexion/extension, internal/external rotation, varus/valgus, anterior/posterior translation, medial/lateral translation, proximal/distal translation.
Kinematic characteristics of the 6DOF of the gait at the mid-stance phase in asymptomatic participants and patients with knee osteoarthritis. | 1 Day
  The 6DOF include flexion/extension, internal/external rotation, varus/valgus, anterior/posterior translation, medial/lateral translation, proximal/distal translation.
Kinematic characteristics of the 6DOF of the gait at the maximum motion in swing phase in asymptomatic participants and patients with knee osteoarthritis. | 1 Day
  The 6DOF include flexion/extension, internal/external rotation, varus/valgus, anterior/posterior translation, medial/lateral translation, proximal/distal translation.

SECONDARY OUTCOMES:
Kellgren-Lawrence Scores in patients with knee osteoarthritis. | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zhang, PhD, Study Chair — Hospital of Orthopedics, Guangzhou General Hospital of Guangzhou Military Command, 111 Liuhua Road, Guangzhou 510010, China
Locations (1):
- Hospital of Orthopedics, Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No